CLINICAL TRIAL: NCT00066469
Title: Phase II Study of Cyclophosphamide, Prednisone and Rituximab (CPR) in Children, Adolescents and Young Adults With B-lymphocyte Antigen CD20 (CD20) Positive Post-Transplant Lymphoproliferative Disease (PTLD) Following Solid Organ Transplantation (SOT)
Brief Title: Cyclophosphamide, Rituximab, and Either Prednisone or Methylprednisolone in Treating Patients With Lymphoproliferative Disease After Solid Organ Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANHL0221; CDR0000316241 (Other: Clinical Trials.gov); COG-ANHL0221 (Other: Children's Oncology Group); NCI-2012-02544 (Other: NCI); U10CA098543 (NIH)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Results first posted 2014-01-17 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2016-09

CONDITIONS: Lymphoproliferative Disorder
Keywords: post-transplant lymphoproliferative disorder
MeSH Terms: conditions — Lymphoproliferative Disorders | interventions — Rituximab; Cyclophosphamide; Methylprednisolone; Prednisone; prednisolone phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide, prednisone, rituximab (Experimental): Patients receive cyclophosphamide IV over 30-60 minutes on day 1 and oral prednisone or methylprednisolone IV twice daily on days 1-5. During courses 1 and 2 only, patients also receive rituximab IV over 2-5 hours on days 1, 8, and 15. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression, a new primary or secondary malignancy, or unrelated disease
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: methylprednisolone; Drug: prednisone

INTERVENTIONS:
Biological: rituximab — Cycles 1 and 2 only: Given IV Incremental: First dosage: < 21 years of age: 0.5mg/kg/hr (maximum of 50 mg/hr) for the 1st hour ≥ 21 years of age: 50 mg/hr for the 1st hour. Subsequent dosages: < 21 years of age: 1.0mg/kg/hr (maximum of 50 mg/hr) for the 1st hour ≥ 21 years of age: 100 mg/hr for the 1st hour. Days 1, 8 and 15.
  Other Names: IDEC-C2B8; NSC #687451
Drug: cyclophosphamide — Given IV over 30-60 minutes Dose 600 mg/m2 in 50-250 mL of normal saline (NS) or Dextrose-Water 5%(D5W) (at a maximum concentration of 20 mg/ml) over 30-60 minutes on day 1 of each cycle
  Other Names: Cytoxan; NSC #26271
Drug: methylprednisolone — Methylprednisolone 0.8 mg/kg IV over 12 hours on days 1,2,3,4 and 5 of each cycle.
  Other Names: Deltaone; Meticorten; Orasone; Liquid Pred; Pediapred; Sterapred; NSC #010023
Drug: prednisone — Dosage 1 mg/kg orally every 12 hours on days 1,2,3,4 and 5 of each cycle. Oral prednisone may be rounded up to the nearest 2.5 mg as necessary for tablet size
  Other Names: Deltaone; Meticorten; Orasone; Liquid Pred; Pediapred; Sterapred; NSC #010023

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as cyclophosphamide, prednisone, and methylprednisolone use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining cyclophosphamide and either prednisone or methylprednisolone with rituximab may be effective in treating lymphoproliferative disease following organ transplantation.

PURPOSE: Phase II trial to study the effectiveness of combining cyclophosphamide and either prednisone or methylprednisolone with rituximab in treating patients who have Epstein-Barr virus-positive lymphoproliferative disease following organ transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of cyclophosphamide, rituximab, and prednisone or methylprednisolone in patients with CD20-positive and Epstein-Barr virus-positive post-transplant lymphoproliferative disease (PTLD) after solid organ transplantation.
* Determine the 2-year event-free survival, defined as alive and in continuous complete remission with a functioning original allograft, of patients treated with this regimen.
* Determine the response rate in patients treated with this regimen.
* Determine the PTLD gene expression profile by microarray analysis and fluorescent in situ hybridization in patients treated with this regimen.
* Determine the accrual rate of patients to this study.

OUTLINE: This is a multicenter study.

Patients receive cyclophosphamide IV over 30-60 minutes on day 1 and oral prednisone or methylprednisolone IV twice daily on days 1-5. During courses 1 and 2 only, patients also receive rituximab IV over 2-5 hours on days 1, 8, and 15. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression, a new primary or secondary malignancy, or unrelated disease.

After finishing study treatment, patients are followed periodically for at least 5 years.

PROJECTED ACCRUAL: A total of 60 patients (50 with non-fulminant post-transplant lymphoproliferative disease [PTLD] and 10 fulminant PTLD) will be accrued for this study within 2.5-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed post-transplant lymphoproliferative disease (PTLD)

  * Presents with 1 of the following:

    * Fulminant PTLD (F-PTLD)

      * Fever greater than 38°C
      * Hypotensive (for age)
      * Evidence of multiple organ involvement/failure, including at least 2 of the following:

        * Marrow (including pancytopenia without detectable B-cell proliferation)
        * Liver (coagulopathy, transaminitis, and/or hyperbilirubinemia)
        * Lungs (interstitial pneumonitis with or without pleural effusions)
        * Gastrointestinal tract hemorrhage
    * Non-fulminant PTLD (NF-PTLD)

      * Does not meet the above F-PTLD criteria
      * Considered medically refractory to reduced immune suppression (50% or more reduction of immunosuppression) for at least 1 week
* CD20 positive AND Epstein-Barr virus positive
* Must have received prior solid organ transplantation
* Must have residual disease after biopsy and/or surgery
* No PTLD central nervous system (CNS) disease, defined as positive cytology and/or radiographic evidence

PATIENT CHARACTERISTICS:

Age

* Under 31

Performance status

* Not specified

Life expectancy

* NF-PTLD patients:

  * At least 8 weeks

Hematopoietic

* See Disease Characteristics

Hepatic

* See Disease Characteristics

Renal

* Not specified

Pulmonary

* See Disease Characteristics

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 1 month since prior rituximab

Chemotherapy

* More than 4 weeks since prior chemotherapy and recovered

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2004-04; Primary Completion 2009-10-01 (Actual); Study Completion 2013-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Gross, MD, PhD, Study Chair — Nationwide Children's Hospital
Locations (78):
- United States (66):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Illinois Cancer Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- Australia (3):
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (7):
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
- New Zealand (2):
  - Starship Children's Health, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- [Result] Gross TG, Orjuela MA, Perkins SL, Park JR, Lynch JC, Cairo MS, Smith LM, Hayashi RJ. Low-dose chemotherapy and rituximab for posttransplant lymphoproliferative disease (PTLD): a Children's Oncology Group Report. Am J Transplant. 2012 Nov;12(11):3069-75. doi: 10.1111/j.1600-6143.2012.04206.x. Epub 2012 Aug 6. PMID 22883417

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyclophosphamide, Prednisone, Rituximab
Started | 55
Completed | 39
Not Completed | 16
Not completed — Death | 3
Not completed — Lack of Efficacy | 9
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide, Prednisone, Rituximab
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 38
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 46
  Canada | 7
  Australia | 2

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Alive in continuous complete remission with functioning original allograft. The Event Free Survival (EFS) will be estimated by the Kaplan-Meier method.
Time Frame: 2 years
Population: One patient out of the 55 patients enrolled was ineligible for study and therefore was excluded from analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants analyzed
Arm/Group | Cyclophosphamide, Prednisone, Rituximab
Number analyzed (Participants) | 54
percentage of participants analyzed | 71 [57 to 82]

ADVERSE EVENTS:
Description: One patient out of the 55 patients enrolled was not eligible for this study. Only eligible patients were included in the Adverse Event (AE) analysis for both Serious and Other AE events.
Arm/Group | Cyclophosphamide, Prednisone, Rituximab
Serious Adverse Events (participants affected / at risk) | 2/54
Other Adverse Events (participants affected / at risk) | 38/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide, Prednisone, Rituximab (N=54)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide, Prednisone, Rituximab (N=54)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (12)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 3 (3)
Enterocolitis infectious (Infections and infestations) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 17 (17)
Kidney infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Peritoneal infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Small intestine infection (Infections and infestations) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Blood bilirubin increased (Investigations) | 3 (3)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 4 (4)
GGT increased (Investigations) | 5 (5)
Investigations - Other, specify (Investigations) | 1 (1)
Lipase increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 15 (15)
Platelet count decreased (Investigations) | 2 (2)
Serum amylase increased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 9 (9)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (6)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1)
Renal hemorrhage (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.